CLINICAL TRIAL: NCT07038642
Title: The Electronic Asthma Management System in Pharmacies (eAMS-Pharm)
Brief Title: The Electronic Asthma Management System in Pharmacies
Acronym: eAMS-Pharm
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Samir Gupta, Clinician Scientist, Unity Health Toronto
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 46441
Record Dates: First submitted 2025-06-05; First posted 2025-06-26 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Pharmacy; Asthma Management; Asthma; Computerized Decision Support System
Keywords: Asthma; Pharmacy; Asthma management; Computerized decision support system
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Interrupted time series analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control - None (No Intervention): A retrospective, pharmacy chart review will assess pharmacy-delivered care in the six-month pre-intervention period.
- Intervention - The Electronic Asthma Management System in Pharmacies (eAMS-Pharm) (Active Comparator): Throughout the intervention period, the eAMS-Pharm will be provided to pharmacists/RPhTs/assistants/students (for use in eligible patients).
  Interventions: Behavioral: Pharmacy Clinical Decision Support System for Asthma Management

INTERVENTIONS:
Behavioral: Pharmacy Clinical Decision Support System for Asthma Management — A pharmacy clinical decision support system that generates individualized advice for asthma patients is provided to the pharmacist/RPht/assistant/student.
  Arms: Intervention - The Electronic Asthma Management System in Pharmacies (eAMS-Pharm)

SUMMARY:
The goal of this study is to assess the effect of an electronic asthma management system in pharmacies (eAMS-Pharm) on asthma control assessment, asthma medication adjustment, asthma action plan delivery, and prompting for specialist referral in severe asthma. The study assesses the differences on pharmacy processes (affecting both the pharmacy team and patients) and pharmacy-delivered care using an interrupted time-series analysis (six-months before vs. six-months after the introduction of eAMS-Pharm in study pharmacy sites).

The eAMS-Pharm uses patient data (asthma control, asthma flare-up risk, and current medications) to provide clinical decision support to pharmacists, empowering them to bridge existing gaps between guideline-recommended asthma care and patient care received.

DETAILED DESCRIPTION:
Asthma is the third most common chronic disease in adults and is increasing in prevalence. Although effective therapies exist and well-controlled asthma is achievable in most patients, studies demonstrate that up to 90% of Canadians with asthma are poorly controlled. This poor control and associated health system burden are attributable to 4 major gaps in care: 1) failure to ascertain asthma control according to guideline criteria; 2) failure to escalate pharmacotherapy in response to suboptimal control; 3) failure to provide a written asthma action plan (AAP) (a personalized plan produced by a health care professional for a patient, providing education and guidance for self-management of flares); and 4) failure to refer patients with severe asthma to specialty care for biologic therapies (these were 4 of the 6 quality statements in Health Quality Ontario's Asthma Quality Standards).

The Electronic Asthma Management System (eAMS) is a validated tool that has the potential to address the 4 major gaps in care. The eAMS consists of a web-based portal-based e-questionnaire, which collects asthma parameters directly from patients. A point-of-care Computerized Decision Support System (CDSS) receives and processes questionnaire data to produce guideline-based decision support such as assessments of asthma control, relevant medication change recommendations, and a personalized asthma action plan (AAP). There are also web-based education resources in the patient portal. The eAMS was proven to improve asthma management in primary care across these care gaps and is used in 16 primary care clinics, with ~215 providers and ~7200 patients with asthma. Now, with the increasingly critical role that pharmacists are playing in Canada's healthcare ecosystem, the eAMS can also be used to empower pharmacists to help optimize chronic disease care.

Pharmacists' scope of practice is growing rapidly in Ontario and across Canada. At the same time, asthma control remains suboptimal for millions of Canadians. Furthermore, the eAMS has been extensively studied and validated as an optimal tool to improve asthma management in primary care. The use of the eAMS in pharmacies presents a unique opportunity to involve pharmacists in chronic disease care while also reducing the burden on primary care. To address limited primary care access and given rapid the expansion of pharmacists' role of in care delivery, the investigators adapted the platform to build the eAMS-Pharm - a chronic disease quality improvement tool for pharmacists. The results of this study will inform the broader implementation of the eAMS across pharmacies and similar knowledge translation tools in pharmacies in the future.

ELIGIBILITY:
* Eligible patients would be those who have asthma and are seen at one of the three study pharmacies during the study period
* Eligible pharmacy team members would be staff (pharmacists/RPhTs/assistants/students) at any one of the three study pharmacies

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2025-12-23 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Medication adjustments | 12 months, broken into individual time series periods
  Using pharmacist chart review, the investigators will assess the proportion and trend in patients receiving medication adjustments
Asthma control assessment | 12 months, broken into individual time series periods
  Using pharmacist chart review, the investigators will assess the proportion and trend of patients receiving asthma control assessment by guideline criteria
Asthma action plan creation | 12 months, broken into individual time series periods
  Using pharmacist chart review, the investigators will assess the proportion and trend of asthma action plans being created for patients

SECONDARY OUTCOMES:
System usage: virtual and in-person visit frequency | 6 months
  Using pharmacist chart review, investigators will assess the number of times the system was used in virtual (i.e., telemedicine) visits and in in-person visits
System usage: content access frequency | 6 months
  Using system analytics, investigators will assess the type of content accessed (clinical tools, clinical decisions, educational materials) by patients and pharmacy teams
System usage: patient engagement frequency, by method | 6 months
  Using system analytics, investigators will assess the number of patients who engaged with the system by the programmatic (mass invite) method, or as a walk-in patient following programmatic invitations
System usage: time required for access and documentation | 6 months
  Using system analytics, investigators will assess how long it takes pharmacy teams to access and complete clinical decision making within the system. Last screen timestamp minus first screen timestamp will be used to measure time
Quantitative patient Likert-Scale questionnaire | 6 months
  Exclusively throughout the intervention, electronic questionnaires developed by the investigators will be sent to consenting patients to assess quantitative patient feedback on system functionality and care quality received, as 5-point Likert scales. Multiple choice and yes/no questions will also bee used to determine demographics and relevant asthma diagnosis information
Qualitative patient free-text feedback questionnaire | 6 months
  Exclusively throughout the intervention, electronic questionnaires developed by the investigators will be sent to consenting patients to assess qualitative patient feedback on benefits and drawbacks of the system, as measured through two free-text questions
Pharmacy team feedback: 10-item System Usability Scale - SUS | 6 months
  Exclusively throughout the intervention, electronic questionnaires developed by the investigators will be sent to consenting pharmacy team members to assess feedback on system usability, as measured by The System Usability Scale (SUS), a 10-item 5-point Likert scale
Quantitative pharmacy Likert-Scale questionnaire | 6 months
  Exclusively throughout the intervention, electronic questionnaires developed by the investigators will be sent to consenting pharmacy team members to assess quantitative pharmacy team feedback on technology interest, role of pharmacies in chronic disease care and asthma action plans, system functionality, and benefits and drawbacks of the system on pharmacy workflows, as measured with 5-point Likert scales
Qualitative pharmacy free-text feedback questionnaire | 6 months
  Exclusively throughout the intervention, electronic questionnaires developed by the investigators will be sent to consenting pharmacy team members to assess qualitative pharmacy team feedback on system usage, as measured through 6 free text questions. To supplement the outcome of revenue metrics, the pharmacy team feedback questionnaire will also ask pharmacy team members to estimate revenue for time spent
Prescription/action plan sign-back proportions | 12 months, broken into individual time series periods
  Using pharmacist chart review, the investigators will assess the proportion of prescriptions/action plans which receive sign-back from prescribers in each analysis period
Revenue metrics: pharmaceutical opinion proportion | 12 months, broken into individual time series periods
  Using pharmacist chart review, the investigators will assess the proportion of eligible visits for which a pharmaceutical opinion was successfully billed
Revenue metrics: MedsCheck proportion | 12 months, broken into individual time series periods
  Using pharmacist chart review, the investigators will assess the proportion of eligible visits for which a MedsCheck was successfully billed
Revenue metrics: total dollar revenue per patient | 12 months, broken into individual time series periods
  Using pharmacist chart review, the investigators will assess the total average revenue per eligible patient by summing pharmaceutical opinion, MedsChecks, markups, and dispensing fees
Revenue metrics: dollar reimbursement for time spent in system | 6 months
  Using pharmacist chart review, the investigators will assess the overall reimbursement for time pharmacy team members spent in the system. To measure, investigators will sum the total revenue per patient and divide by time spent in the system for each patient over visits. An average will be calculated across all patients
Specialist referral prompt proportion | 12 months, broken into individual time series periods
  Using pharmacist chart review, the investigators will assess the proportion of severe asthma patients, as identified by medications currently prescribed and filled, and who are not already seeing a specialist, for whom a prompt for specialist referral was sent to the prescriber

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Medical Place Pharmacy, Ajax, Ontario
  - LiveWell Pharmacy, Niagara Falls, Ontario
  - Westmount Place Pharmacy, Waterloo, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: eAMS-Pharm web page — https://easthma.ca/pharmacists